CLINICAL TRIAL: NCT02755779
Title: Characterization of Breast Masses Incidentally Detected on Chest CT - a Prospective Study
Brief Title: Characterization of Breast Masses Incidentally Detected on Chest CT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Yoav Amitai, Dr, Tel Aviv Medical Center
Other Study IDs: 0067-16-TLV
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Although Computed tomography (CT) is not routinely used to evaluate beast masses, It is common to discover Incidental breast lesions on chest CT.

The goal of this study is to investigate the incidence and appearance of incidentally discovered breast masses on chest CT.

ELIGIBILITY:
Inclusion Criteria:

* Woman with incidentally discovered breast masses on chest CT

Exclusion Criteria:

* Male gender
* Known breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Woman over 18
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Patient enrollment | One year
  Enrolling 100 patients with breast masses to study

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Amitai, Dr, Principal Investigator — Sourasky medical center Tel aviv

IPD SHARING:
Plan to Share IPD: No